CLINICAL TRIAL: NCT03899727
Title: Sleep Disturbance in Pregnant Women in Upper Egypt
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: SDUE
Record Dates: First submitted 2019-04-01; First posted 2019-04-02 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant group: pregnant women in the third trimester of pregnancy
  Interventions: Device: Polysomnography
- Non-pregnant group: middle aged women
  Interventions: Device: Polysomnography

INTERVENTIONS:
Device: Polysomnography — Polysomnography, also called a sleep study, is a test used to diagnose sleep disorders. Polysomnography records your brain waves, the oxygen level in your blood, heart rate and breathing, as well as eye and leg movements during the study

SUMMARY:
Pregnant women are associated with hormonal, anatomic and mechanical changes that Change sleep patterns and quality of sleep. Several Investigators have reported Associations between sleep disturbances and hypertension, Coronary artery disease, Diabetes, and depression. Most of these associations have been established in the association with sleep disturbances

ELIGIBILITY:
Inclusion Criteria:

* All viable third trimester pregnancy

Exclusion Criteria:

* Intrauterine fetal death
* Any History of neurological, mental disorder.
* Any previous diagnosed sleep disturbances breathing disorder before pregnancy.
* Any patient with respiratory infection in the pregnancy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients visiting out patient clinic at Women Health Hospital will be counseled to participate in our study careful history taking and examination to exclude patients who not eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
The percentage of women with sleep disturbances among overall included women | 30 minutes
  diagnosis of sleep disturbances will depend on STOP and STOP-Bang questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No